CLINICAL TRIAL: NCT02313012
Title: A Phase 1a Multicenter, Open-label Safety, Tolerability and Pharmacokinetic Study of CC-90003, a Selective Extracellular Signal-Regulated Kinase (ERK) Inhibitor, in Subjects With Locally-Advanced or Metastatic, Relapsed, or Refractory BRAF or RAS-Mutated Malignancies
Brief Title: Safety and PK Study of CC-90003 in Relapsed/Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90003-ST-001
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Neoplasm Metastasis
Keywords: Maximum Tolerated Dose; Solid Tumors; Locally Advanced Tumors; Metastatic Solid Tumors; Relapsed or refractory, BRAFV600 or RAS-mutated solid tumors; Melanoma; Colorectal Carcinomas Papillary; Thyroid carcinomas; Pancreatic ductal Adenocarcinomas; Non -small cell lung cancer [NSCLC]
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Melanoma; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Level 1 CC-90003 (Experimental): CC-90003 by mouth (PO) daily on days 1 -21 of every 28 day cycle; Cycle 1, Days 1 to 28 will constitute the dose limiting toxicity (DLT) assessment period for purposes of non-tolerated dose (NTD) and Maximum Tolerated Dose determination.
  Interventions: Drug: CC-90003

INTERVENTIONS:
Drug: CC-90003 — CC-90003 PO once daily

SUMMARY:
The CC-90003-ST -001 trial is a first-in-man, open-label study in subjects with locally-advanced or wide spread cancers to determine if CC-90003 (an oral medication) can be adequately tolerated with minimal side effects.

DETAILED DESCRIPTION:
CC-90003-ST -001 is an open-label, multicenter, Phase 1a study in subjects with locally-advanced or metastatic, solid tumors who are intolerant of, resistant to, or have relapsed after at least one line of therapy and for whom no standard therapy exists. The study will be conducted in two parts: Dose Escalation (Part 1) and Cohort Expansion (Part 2). Subjects may continue CC-90003 until progression of their underlying malignancy, the occurrence of intolerable toxicity, or physician/subject decision to discontinue CC-90003. In Part 1, cohorts of subjects with relapsed or refractory solid tumors will receive increasing doses of CC-90003 in order to assess its safety and tolerability, the maximum tolerated dose (MTD), and PK profile. In Part 2, cohorts of subjects with specific tumors that harbor mutations involving the Mitogen -Activated Protein Kinase (MAPK) pathway will receive CC-90003 at or below the MTD until progression of disease, intolerable toxicity, or physician/subject decision to discontinue CC-90003.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible study subjects in Part 1 and Part 2 must be 18 years or older
2. Eligible study subjects must have histologic or cytologic confirmation of advanced, unresectable or metastatic solid tumors, and have at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
3. Eligible study subjects must have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
4. Eligible study subjects must exhibit acceptable liver, bone marrow, renal and cardiac functions as assessed by laboratory tests, ECG and ECHO or MUGA scan.

Exclusion Criteria:

1. Subjects with symptomatic or unstable CNS metastases
2. Subjects with a history of recent (within 28 days) systemic therapy for their underlying malignancy
3. Subjects who have had surgery/radiotherapy within 2 weeks prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-03 (Actual)

PRIMARY OUTCOMES:
Summary of the adverse events (type, severity, and incidence) related to CC- | Up to 36 months
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values regardless of etiology.
Dose Limiting Toxicities of CC-90003 | Up to 18 months
  Number of participants with dose limiting toxicities during the Dose Escalation Phase
Maximum Tolerated Dose (MTD) of CC-90003 | Up to 36 months
  The MTD is defined as the highest dose level at which no more than 1 in 6 participants experiences a dose- limiting toxicity (DLT) during the first 28 day cycle of treatment
Pharmacokinetics (PK) observed maximum concentration (Cmax) | Cycle 1, Day 1, 2, 3 (predose), 8, 11 (predose), 15, 16, , Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  The maximally observed plasma concentration of CC-90003 (Cmax)
PK-Area under the plasma concentration time curve (AUC) | Cycle 1, Day 1, 2, 3, (predose) 8, 11 (predose), 15, 16, Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  Area under the plasma concentration -time curve of CC-90003
PK-Time to maximal plasma concentration (Tmax) | Cycle 1, Day 1, 2, 3 (predose) 8, 11 (predose), 15, 16, Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  The time to reach Cmax
PK- terminal half-life; t1/2 | Cycle 1, Day 1, 2, 3 (predose) 8, 11 (predose), 15, 16, Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  Terminal phase elimination half-life (t1/2) is calculated as follows: t1/2 =ln(2)/λz, where λz is the first order rate constant associated with the terminal portion of the CC-90003 plasma concentration curve
PK-Apparent total body clearance (CL/F) | Cycle 1, Day 1, 2, 3 (predose) 8, 11 (predose) 15, 16, , Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  The apparent total body clearance of CC-90003 from plasma
PK- Apparent Total Volume of Distribution (Vz/F) | Cycle 1, Day 1, 2, 3 (predose) 8, 11 (predose), 15,16, Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  PK- Apparent Total Volume of Distribution (Vz/F) During the terminal phase for CC- 90003
Accumulation index of CC-90003 | Cycle 1, Day 1, 2, 3 (predose) 8, 11 (predose), 15, 16, Cycle 2, Day 1, Cycle 3, Day 1 and at discontinuation
  Accumulation represents the relationship between the dosing interval and the rate of elimination for the drug

SECONDARY OUTCOMES:
Response Rate based on RECIST 1.1 | Up to 36 months
  The proportion of subjects who achieve a best response of CR or PR.
Duration of Response | Up to 36 months
  Duration of response is the time from the start of study treatment until the first documentation of an objective response (either CR or PR).
Disease Control | Up to 36 Months
  The proportion of subjects who achieve a best response of SD (documented at least 56 days after the start of study treatment) PR, or CR
Progression Free Survival | Up to 36 months
  PFS is defined as the time from the start of study treatment until progression (PD) or patient death (any cause), whichever occurs first
Overall Survival | Up to 36 months
  Overall survival is defined as the time from start of study treatment until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bray, MD, Study Director — Celgene
Locations (5):
- United States (4):
  - Cedars Sinai Medical Center, Inflammatory Bowel Disease Center, Los Angeles, California
  - Smilow Cancer Center, New Haven, Connecticut
  - Levine Cancer Institute, Charlotte, North Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
- Peter MacCallum Cancer Centre, Melbourne, Australia